CLINICAL TRIAL: NCT05285111
Title: Pilot of Reconnecting to Internal Sensations and Experiences in Undergraduates
Acronym: RISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, April Smith, Assistant Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-001
Record Dates: First submitted 2022-02-01; First posted 2022-03-17 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Suicidal Ideation; Eating Disorder Symptom
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interoceptive Awareness (Experimental): The intervention consists of four modules that focus on multiple aspects of interoception including: body awareness, body sensations/movement, eating, health and self-care, emotional awareness, and understanding the self in relation to others.
  Interventions: Behavioral: Reconnecting to Internal Sensations and Experiences
- Healthy Habits (Active Comparator): The comparator condition is called "Health Habits" and is matched for time and attention; participants complete modules related to healthy habits such as financial planning, hygiene, stretching, and healthy eating.
  Interventions: Behavioral: Healthy Habits

INTERVENTIONS:
Behavioral: Reconnecting to Internal Sensations and Experiences — The intervention consists of four modules that focus on multiple aspects of interoception including: body awareness, body sensations/movement, eating, health and self-care, emotional awareness, and understanding the self in relation to others.
  Arms: Interoceptive Awareness
Behavioral: Healthy Habits — The comparator condition is called "Health Habits" and is matched for time and attention; participants complete modules related to healthy habits such as financial planning, hygiene, stretching, and healthy eating.
  Arms: Healthy Habits

SUMMARY:
Project RISE is a randomized control trial. The intervention consists of four modules that focus on multiple aspects of interoception including: body awareness, body sensations/movement, eating, health and self-care, emotional awareness, and understanding the self in relation to others. The comparator condition is called "Health Habits" and is matched for time and attention; participants complete modules related to healthy habits such as financial planning, hygiene, stretching, and healthy eating. Variables of interest include self-report measures of interoception, eating pathology, suicidality, physiological measures of interoception (electrocardiograph; ECG; pain tolerance measured via algometer), and an implicit association test (IAT) with death and life stimuli (meant to measure implicit associations with suicidality). The population will be college students, with current or past suicidality or low interoception.

ELIGIBILITY:
Inclusion Criteria:

* Low interoceptive awareness
* History of suicidal ideation or attempt
* 18 or older

Exclusion Criteria:

*Below the age of 18

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Multidimensional Assessment of Interoceptive Awareness | within one week of Post-test
  Assessment of Interoceptive Awareness. Total scores range from 0-175. Higher scores indicate a better outcome.
Treatment acceptability | within one week of Post-test
  Feasibility and Acceptability questions. Scores range from 4-28. Higher scores indicate a better outcome.

SECONDARY OUTCOMES:
Depression Screening Inventory-Suicidality Subscale | within one week of Post-test
  Measure of suicidal ideation, greater scores indicate more severe ideation. Scores range from 0-12. Higher scores indicate more suicidality, or a worse outcome.
Eating Disorder Examination Questionnaire | within one week of Post-test
  Measure of disordered eating. Global score ranges from 0-6; greater scores indicate more severe eating disorder symptoms
Heartbeat perception task | within one week of Post-test
  Measured via ECG. Perceived versus actual heartbeats are recorded across 3 trials. Scores range from 0-1; higher scores indicate greater cardiac interoceptive accuracy.
Brief Symptom Inventory | within one week of Post-test
  Short measure assessing anxiety and depression symptoms. Scores range from 0-72; greater scores indicate more pathology

CONTACTS AND LOCATIONS:
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No